CLINICAL TRIAL: NCT02136953
Title: An Examination of Structured Physical Exercise in OCD: Treatment Efficacy, Additive Benefits to CBT, and Cognitive Correlates of Change
Brief Title: Physical Exercise in OCD: Treatment Efficacy, Additive Benefits to CBT, and Cognitive Correlates of Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre for Addiction and Mental Health (Other); McMaster University (Other); Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr. Neil Rector, Research Scientist, Psychologist, and Director of the Mood and Anxiety Treatment and Research Program, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MOP133452
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Obsessive-Compulsive Disorder; Cognition Disorders
Keywords: Obsessive-Compulsive Disorder; Exercise; Cognitive Behavior Therapy; Cognitive Behavioral Therapy; Treatment Efficacy; Brain-Derived Neurotrophic Factor
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Cognition Disorders; Motor Activity | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Exercise (Experimental): 12-weeks of structured, individual aerobic exercise, 3 times a week, increasing from 15-30 minutes to 30-40 minutes per session.
  Interventions: Behavioral: Exercise
- Cognitive Behavioural Therapy (CBT) (Active Comparator): 12-weeks of manual-based group CBT, 2 hours per week, 8 participants per group.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)
- Exercise and CBT (Experimental): Combined 12-week Exercise program and CBT.
  Interventions: Behavioral: Exercise; Behavioral: Cognitive Behavioural Therapy (CBT)
- Waitlist Condition (No Intervention): 12-week waitlist control condition, after which participants will have the chance to receive CBT group treatment.

INTERVENTIONS:
Behavioral: Exercise — 12 weeks of structured aerobic exercise, 3 times a week, following a two-stage graduated regimen: 1) Initial stage (weeks 1-4): 40-60% intensity, 15-30 min duration (+ 5 min warm-up/cool-down), and 2) Improvement stage (weeks 5-12): 60-80% intensity, 30-45 min duration. Adherence measures include self-reported exercise session logs and weekly phone checks by research assistants.
  Arms: Exercise; Exercise and CBT
Behavioral: Cognitive Behavioural Therapy (CBT) — CBT will be delivered in group format, 2 hours per week, for 12 consecutive weeks with 8-10 participants per group and will be conducted according to a session-by-session treatment manual that incorporates Exposure and Response Prevention (ERP) in the early phases of treatment and then increases emphasis on cognitive approaches for obsessions and compulsions outlined in step-by-step strategies.
  Arms: Cognitive Behavioural Therapy (CBT); Exercise and CBT

SUMMARY:
Obsessive compulsive disorder (OCD) is a severe and debilitating anxiety disorder afflicting 2% of the population. Cognitive behavioural therapy (CBT) is considered first line psychological treatment for OCD, but there are a large number of treatment non-responders, and the majority of responders have residual symptoms. Aerobic exercise has shown potential benefit for general mood and anxiety disorders, but has not been widely tested in OCD. This study will examine the additive benefits of a standard 12-week aerobic exercise program to a standard 12-week CBT protocol in the treatment of OCD. The study will test if Exercise+CBT results in significantly better clinical outcomes compared to either treatment alone or no treatment at all. Treatment outcomes will be assessed in relation to symptom and cognitive measures of clinical improvement.

DETAILED DESCRIPTION:
This study aims to determine if a standard, evidence-based 12-week aerobic exercise program results in significant reduction of obsessive-compulsive symptom severity and associated cognitive dysfunction as a stand-alone intervention and when combined with the first-line psychological treatment, cognitive behavioural therapy (CBT). There are 3 broad aims to this study: 1) to compare the relative efficacy of Exercise, CBT, and their combination (CBT+Ex) versus a non-treatment waitlist control (WL), 2) to examine the extent to which neuropsychological features of OCD improve following treatments, and 3) to determine the extent to which the BDNF gene and protein are a) associated with learning and cognitive factors, and b) moderate symptom and cognitive change across treatments.

The study design allows for a novel, well-powered and potentially landmark study on the impact of exercise on obsessive-compulsive symptom severity and cognitive functioning in OCD, both as a stand-alone treatment and when augmenting CBT. If this study can demonstrate that a short aerobic exercise program of 12 weeks duration can confer significant clinical gains for those suffering with OCD, then it could easily be translated into highly accessible, routine clinical care. Further, demonstration of improvement in OCD-associated cognitive dysfunction, given the refractory nature of the illness, would provide another avenue into the long-term enhancement of outcomes for this chronically affected population.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with DSM-5 diagnosed OCD
* Score of >16 on the Yale-Brown Obsessive Compulsive Scale (YBOCS)
* A Physical Activity Readiness Questionnaire (PAR-Q) score of ≤1
* If on medications for OCD, must be stabilized, i.e. are currently receiving an adequate dose (equivalent of 40mg/day of fluoxetine) for an adequate duration (at least 12 weeks of treatment) prior to the initiation of the study
* Has physician letter of approval for safe participation in fitness assessment and exercise protocol

Exclusion Criteria:

* Previous course of CBT treatment (≥ 8 sessions) in past two years
* Engaging in an active exercise regimen (>2 days/wk of moderate-to-vigorous exercise training) at the time of recruitment
* Concurrent diagnosis of a severe mood disorder, schizophrenia or other psychotic disorders, or substance abuse/dependence
* Suspected organic pathology
* Active comorbid medical condition that may require urgent intervention during the treatment
* Incapable of providing informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in OCD symptom severity, as measured by the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Baseline and 12 weeks
  OCD symptom severity will be measured using the Yale-Brown Obsessive Compulsive Scale (YBOCS).The YBOCS is a standardized rating scale measuring 10 items pertaining to obsessions and compulsions on a 5-point Likert scale ranging from 0 (no symptoms) to 4 (severe symptoms). Both the self-report and clinician interview versions of the YBOCS have been shown to possess high internal consistency and validity.

SECONDARY OUTCOMES:
Change from baseline in cognitive domains sensitive to OCD, as measured by a targeted neuropsychological battery | Baseline to 12 weeks
  We have included core paper-and-pencil and computerized tests, such as those from the Cambridge Neuropsychological Test Automated Battery (CANTAB), which tap separable cognitive domains that are sensitive to OCD. CANTAB measures are standardized and have been shown to discriminate amongst many neurological and psychiatric illnesses To avoid practice effects, measures were selected to have either alternate form or to be amenable to calculation of reliable change indices (RCIs). RCIs will be used to determine if neuropsychology performance scores change significantly over time.

OTHER OUTCOMES:
Change from baseline in fitness level as measured by incremental maximal exercise test | Baseline to 12 weeks
  Participants will undergo an incremental maximal exercise test on an electronically braked cycle ergometer (Lode Corival) to establish level of fitness. Peak heart-rate, peak watts, total duration and ratings of perceived exertion are all recorded during the test. Peak heart-rate will also be used to tailor the aerobic Exercise treatment to the individual participant in order to maximize health benefit.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - St. Joseph's Healthcare Hamilton at McMaster University, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario